CLINICAL TRIAL: NCT07032259
Title: Regenerative Outcomes for Peri-implant Bony Defects Using Amnion-chorion Barrier vs. Collagen Membrane: a Randomized Controlled Clinical Trial
Brief Title: Regenerative Outcomes for Peri-implant Bony Defects Using Amnion-chorion Barrier vs. Collagen Membrane
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Maxxeus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5250224
Record Dates: First submitted 2025-06-19; First posted 2025-06-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Peri-Implantitis
Keywords: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Number of Study Arms/Groups:
  The study includes two arms:
  1. Test Group: Patients receiving amnion-chorion membrane (ACM) during GBR treatment.
  2. Control Group: Patients receiving a standard collagen membrane during GBR treatment.
     * Study Center:
  This is a single-center study conducted at Loma Linda University School of Dentistry, Center for Implant Dentistry.
  * Study Agents / Interventions:
    * Test Intervention: Amnion-chorion membrane (ACM) - dehydrated human placental tissue used as a biologically active resorbable barrier.
    * Control Intervention: Collagen membrane - a conventional resorbable membrane used in GBR procedures.
  * Changes in Scheduling or Dosing:
  No dose escalation or multiple dosing is involved. Both membranes are used locally, applied during a single surgical procedure. Follow-up evaluations will occur at 3, 6, 12, 18, and 24 months postoperatively.
Who Masked: Participant, Outcomes Assessor
Masking Description: This means the patient and the evaluator collecting outcome data (probing, PROMs, radiographs) are blinded. The only one that will not be blinded will be the surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amnion Chorion Membrane (Experimental): Participants in this group will undergo guided bone regeneration for peri-implantitis using an amnion-chorion membrane (ACM) as the barrier membrane during surgical treatment.
  Interventions: Device: BioXclude Amnion Chorion Membrane
- Collagen Membrane (Active Comparator): Participants in this group will undergo guided bone regeneration for peri-implantitis using a conventional collagen membrane as the barrier membrane during surgical treatment.
  Interventions: Device: Collagen Membrane

INTERVENTIONS:
Device: BioXclude Amnion Chorion Membrane — A resorbable allograft membrane derived from dehydrated human amnion and chorion tissue. The membrane is placed over peri-implant bony defects during guided bone regeneration to act as a biological barrier and promote tissue healing.
  Other Names: Amnion Chorion Membrane; ACM
  Arms: Amnion Chorion Membrane
Device: Collagen Membrane — A resorbable xenograft membrane derived from porcine collagen. The membrane is placed over peri-implant bony defects during guided bone regeneration to support space maintenance and facilitate bone regeneration.
  Arms: Collagen Membrane

SUMMARY:
The purpose of this study is to compare the clinical and radiographic outcomes of two different barrier membranes-amnion-chorion membranes (ACM) and conventional collagen membranes-used in guided bone regeneration (GBR) procedures for the treatment of peri-implantitis. Both membranes are commonly used in clinical practice; however, this study aims to determine whether ACM offers greater benefits in terms of peri-implant probing depth reduction, radiographic bone fill, and patient-reported post-operative healing outcomes. The findings may help inform surgical decision-making and support the use of ACM as a more effective regenerative material for managing peri-implant bony defects.

DETAILED DESCRIPTION:
Peri-implantitis is a common complication characterized by inflammation and progressive bone loss around dental implants. Guided bone regeneration (GBR) is a frequently employed surgical approach to manage peri-implant defects. Barrier membranes play a critical role in GBR by excluding soft tissue and supporting bone regeneration.

This randomized controlled clinical trial is designed to compare the outcomes of two commonly used barrier membranes: amnion-chorion membranes (ACM) and conventional collagen membranes. Although both are used in practice, ACM may offer additional biological benefits due to the presence of growth factors, anti-inflammatory properties, and native extracellular matrix components.

The study will enroll 56 participants across four clinical sites, with subjects randomly assigned to receive either ACM or a collagen membrane during peri-implant GBR surgery. Clinical parameters, including probing depths and peri-implant soft tissue health, will be recorded at baseline and follow-up visits. Patient-reported outcome measures (PROMs) will be collected using standardized questionnaires to evaluate post-operative healing, discomfort, and satisfaction. Standardized periapical radiographs will be taken at 3, 6, 12, 18, and 24 months to assess radiographic bone fill.

The primary objective is to determine whether the use of ACM results in improved clinical and radiographic outcomes compared to collagen membranes. Secondary objectives include evaluating patient-reported healing and long-term implant stability. Results from this study may inform clinical decision-making and potentially support the wider use of ACM in regenerative peri-implant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adults (≥18 years) with a diagnosed peri-implantitis lesion requiring surgical intervention of any ethnicity
* Comprehension of treatment plan and research project.
* Presence of a single implant in function for at least one year.
* Radiographic evidence of peri-implant bone loss not exceeding one-third of the implant length.
* 2-3 wall defects amenable to guided bone regeneration (GBR).
* Screw-retained, posterior, self-cleansing implant prosthesis.
* Commitment to maintaining oral hygiene and attending follow-up visits.

Exclusion Criteria:

* Patients who have had a history of periodontitis, diabetes, smoking habit, or have been prescribed medications that may interfere with bone healing and metabolism
* Patients with allergies to any treatment devices
* Patients who have a lack of keratinized mucosa (<2 mm), or positioning for implants or restorative designs that compromise oral hygiene
* Peri-implant bone defects not attributable to peri-implantitis (e.g. surgical iatrogenic, trauma)
* Anterior implant restorations (#'s 6-11, #'s 22-27) or cement-retained restorations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Peri-Implant Probing Depths | Baseline, 3, 6, 12, 18, and 24 months post-operatively
  Mean reduction in peri-implant probing depth (in millimeters) measured using a standardized periodontal probe at six time points to assess clinical improvement following guided bone regeneration with either an amnion-chorion or collagen membrane.

SECONDARY OUTCOMES:
Radiographic Bone Fill | Over 2 years
  Assessment of vertical bone fill (in millimeters) around the treated implant sites using standardized periapical radiographs taken at baseline and follow-up visits. Images will be analyzed using calibrated software.
PROMS | Baseline, 3, 6, 12, 18, and 24 months post-operatively
  Patient-reported outcomes will be assessed using a standardized questionnaire evaluating pain, comfort, satisfaction, healing, and communication.
  All items are rated on a 4-point Likert-type scale:
  1 = Poor, 2 = Fair, 3 = Good, 4 = Excellent. Higher scores indicate better outcomes. Two yes/no item captures presence of post-op symptoms (e.g., swelling, bleeding, comfort).

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Lozada, Principal Investigator — Department Chair

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sadowsky SJ. Peri-implantitis after 40 years: Evidence, mechanisms, and implications: A mapping review. J Prosthet Dent. 2024 Dec;132(6):1215-1225. doi: 10.1016/j.prosdent.2023.02.008. Epub 2023 Mar 17. PMID 36935269
- [Result] Monje A, Pons R, Insua A, Nart J, Wang HL, Schwarz F. Morphology and severity of peri-implantitis bone defects. Clin Implant Dent Relat Res. 2019 Aug;21(4):635-643. doi: 10.1111/cid.12791. Epub 2019 May 14. PMID 31087457
- [Result] Baima G, Citterio F, Romandini M, Romano F, Mariani GM, Buduneli N, Aimetti M. Surface decontamination protocols for surgical treatment of peri-implantitis: A systematic review with meta-analysis. Clin Oral Implants Res. 2022 Nov;33(11):1069-1086. doi: 10.1111/clr.13992. Epub 2022 Sep 7. PMID 36017594
- [Result] Bhide VM, Goldberg MB, Tenenbaum HC. Surgical Treatment of Peri-implantitis with Guided Bone Regeneration Using Dehydrated Amnion-Chorion Membranes: A Case Report with a 2-Year Follow-up. Int J Periodontics Restorative Dent. 2022 May-Jun;42(3):e59-e66. doi: 10.11607/prd.5633. PMID 35472107
- [Result] Miller RJ, Korn RJ, Miller RJ. The Use of a Dehydrated, Deepithelialized Amnion-Chorion Membrane in Guided Bone Regeneration Involving Staged Implant Placement: Case Series with a 5-Year Follow-up. Int J Periodontics Restorative Dent. 2021 Sep-Oct;41(5):657-662. doi: 10.11607/prd.5602. PMID 34547066
- [Result] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Clin Periodontol. 2018 Jun;45 Suppl 20:S246-S266. doi: 10.1111/jcpe.12954. PMID 29926484